CLINICAL TRIAL: NCT04651660
Title: Using Electrocochleography to Guide Insertion of the Electrode Array During Cochlear Implantation of the Neuro Zti (eCoN)
Brief Title: Using Electrocochleography During Cochlear Implantation of the Neuro Zti.
Acronym: PIC-22_eCoN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Devices recall due to hermeticity problems.
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIC-22
Record Dates: First submitted 2020-11-19; First posted 2020-12-03 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Cochlear Hearing Loss; Cochlear Trauma
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Insertion (Experimental): The surgeon will follow a classical surgical procedure for the cochlear implantation, i.e. mastoidectomy to access the temporal bone, posterior tympanotomy to access the cochlea and round window (RW) approach for the CI electrode array insertion. Before opening the RW, the eCochG recording electrode is placed on the cochlear promontory, and placed not to obstruct the surgery. The probe is thus maintained during the whole MANUAL insertion (by the surgeon).
  Interventions: Device: Neuro Cochlear Implant System
- Robotic insertion (Experimental): The surgeon will follow a classical surgical procedure for the cochlear implantation, i.e. mastoidectomy to access the temporal bone, posterior tympanotomy to access the cochlea and round window (RW) approach for the CI electrode array insertion. Before opening the RW, the eCochG recording electrode is placed on the cochlear promontory, and placed not to obstruct the surgery. The probe is thus maintained during the whole ROBOTIC insertion.
  Interventions: Device: Neuro Cochlear Implant System

INTERVENTIONS:
Device: Neuro Cochlear Implant System — Before the mastoidectomy, the ear canal is cleaned, the insert earphone is connected to the Eclipse (Oticon Medical software) preamplifier and placed into the ear canal. The EEG scalp electrodes (active, ground electrode) are placed on the patient's head. After the posterior tympanotomy, the reference electrode (eCochG probe) is placed on the cochlear promontory.
  The CI electrode array will be inserted following one of the two possible techniques while the eCochG will be recording. The surgeon will either manually insert the array using the Oticon Medical stylet and following the surgery guides and recommendations from Oticon Medical or will control the Robotol insertion angle and drive the robotic arm in the same way.

SUMMARY:
The main objective of this study is to evaluate the correspondence between eCochG and residual hearing by adding two modifications. First, a novel technique for placing and maintaining the probe in place during the whole insertion will be used. Second, a new metric for estimating the eCochG response will be evaluated (eCochG trauma index). The secondary objective is to find other markers of the cochlear trauma insertion associated to eCochG measures. This will be used to evaluate to which extend a traumatic insertion will be deleterious for the patient's post-operative hearing, and ultimately to prevent trauma to the inner ear. Finally, the potential differences in cochlear trauma resulting of the electrode array insertion from two different surgery techniques will be investigated; Either using a manual insertion or using a robotic arm that will drive the insertion automatically.

DETAILED DESCRIPTION:
Main study procedures and assessments:

* Visit 1 (D-30+/-14) INCLUSION: subject information/consent, inclusion/exclusion criteria, CT-scan, Tonal audiometry
* Visit 2 (D0+/-14) COCHLEAR IMPLANT SURGERY: CT-scan, Intra-op eCochG, eCAP, Impedance
* Visit 3 (D+30+/-14) FOLLOW-UP 1 MONTH: Tonal audiometry, Impedance, Fitting maps
* Visit 4 (D+60+/-14) FOLLOW-UP 2 MONTH: Tonal audiometry, Impedance, Fitting maps, Phonemes
* Visit 5 (D+90+/-14) FOLLOW-UP 3 MONTH: Tonal audiometry, Impedance, Fitting maps, Phonemes

ELIGIBILITY:
Inclusion Criteria:

* > or equal 18 years ;
* Candidate for Neuro Zti EVO cochlear implant system, unilateral or bilateral recipient ;
* Preoperative residual hearing with audiometric thresholds less or equal than 80 dB at 500 Hz, or higher frequencies

Exclusion Criteria:

* Medical or psychological conditions which contraindicate surgery (e.g middle ear infection, tympanic membrane perforation) ;
* Patient with a psychological or linguistic inability to understand the information sheet ;
* Patient under legal protection or deprived of liberty
* Patient included and participating to another trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient between the eCochG trauma index (in µV) and the residual hearing (in dB HL). | Through study completion, an average of 2 years
  The eCochG trauma index correspond to electrophysiological changes of the cochlear response during the CI electrode insertion, and is calculated from the difference between post-insertion and pre-insertion eCochG measure (in µV).
  The hearing loss is calculated from the difference between the post-surgical and pre-surgical hearing thresholds (in dB HL).
  The correspondence is calculated from the correlation coefficient between the eCochG trauma index and the hearing loss.
  It is expected that a potential damage measured by the eCochG during the surgery have affected auditory threshold.

SECONDARY OUTCOMES:
Significant decrease of eCochG trauma index (in µV) for electrode array insertion performed manually compared to robotic. | Through study completion, average of 2 years
  eCochG trauma index (µV) as a result of manual electrode insertion compared with robotic insertion.
  Different behaviors of audiological markers since the cochlea may have suffered from biological cell degradation due to the CI electrode insertion. Allied with cochlear degradation will come increased tissue scar density, subsequently increased resistivity of the biological field to the electrical current. This would imply a cascade effect of electrical and audiological outcomes (higher impedances, higher electrical charges required to evoke a sound or the auditory nerve feedback - eCAP, lower overall performances).
Correlation coefficient between the eCochG trauma index (in µV) and a misplacement of the electrode array inside the cochlea based on CT scan. | Through study completion, average of 2 years
  The misplacement will be quantified with the cochlear coverage (in %) and a subjective assessment of the Eschraghi trauma index for exploratory purpose.
  eCochG trauma index (µV) with placement of the CI electrode array in the cochlea (using Pre and Post surgical CT scans).
Correlation coefficient between the eCochG trauma index (in nV) with the electrical charges (in nC) required to elicit eCAP threshold. | Through study completion, average of 2 years
  eCochG trauma index (µV) with eCAP thresholds (nC).
Correlation coefficient between the eCochG trauma index (in nV) with impedance measurement (in Ω). | Through study completion, average of 2 years
  eCochG trauma index (µV) with CI electrode impedances (Ohm).
Correlation coefficient between the eCochG trauma index (in nV) with fitting map electrical charges (in nC), and slopes of their growth functions. | Through study completion, average of 2 years
  eCochG trauma index (µV) with electrical charge (nC) measured on the patient CI fitting map.
Correlation coefficient between the eCochG trauma index (in nV) with scores of phonemes discrimination (%). | Through study completion, average of 2 years
  eCochG trauma index (µV) with scores (in %) of phonemes recognition.

CONTACTS AND LOCATIONS:
Overall Officials: Yann YN Nguyen, Principal Investigator — Hôpital Pitié-Salpêtrière (Paris)

IPD SHARING:
Plan to Share IPD: No